CLINICAL TRIAL: NCT06008405
Title: Phase Ib Clinical Trial of TQB2928 Injection Combination Therapy in Patients With Hematological Malignancies
Brief Title: Clinical Trial Evaluating the Safety of the TQB2928 Injection Combination Therapy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2928-Ib-01
Record Dates: First submitted 2023-08-18; First posted 2023-08-23 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-03

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Azacitidine; Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2928 Injection + Azacitidine for injection (Experimental): Dose escalation:
  Intravenous infusion of TQB2928 Injection once a week, combined with azacitidine for injection (75 mg/m2, d1-7/q4w), 4 weeks (28 days) as a treatment cycle.
  Dose expansion:
  The maximum tolerated dose (MTD) or optimal biological dose (OBD) or recommended phase II dose (RP2D) determined in the dose-escalation phase is combined with azacitidine for injection for extended studies to further observe the safety and efficacy.
  Interventions: Drug: TQB2928 Injection + Azacitidine for injection

INTERVENTIONS:
Drug: TQB2928 Injection + Azacitidine for injection — TQB2928 injection is a fully humanized Immunoglobulin G 4 (IgG4) subtype monoclonal antibody targeting CD47.
  Azacitidine for injection is a nucleoside metabolism inhibitor that inhibits DeoxyriboNucleic Acid (DNA) methyltransferase, reduces DNA methylation and alters gene expression.

SUMMARY:
This study carried out a phase Ib clinical trial of TQB2928 injection combined therapy in patients with hematological malignancies, to explore the safety, pharmacokinetics, pharmacodynamics and preliminary efficacy of TQB2928 injection combined with azacitidine for injection in Acute Myeloid Leukemia (AML)/Myelodysplastic Syndromes (MDS) subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily join this study, sign the informed consent form, and have good compliance;
* Age: age ≥ 18 years old (when signing the informed consent); Eastern Cooperative Oncology Group Performance Status (ECOG PS) score: 0-2 points; expected survival time of more than 3 months;
* Subject population:

  1. The subjects were diagnosed with AML or MDS according to the World Health Organization (WHO) 2016 revised classification criteria for hematopoietic and lymphoid tissue tumors.
  2. MDS adopts the revised International Prognostic Scoring System (IPSS-R) > 3.5 (higher risk group), and the proportion of bone marrow blasts ≥ 5%.
  3. Phase 1 (dose escalation phase) and Phase 2 (dose expansion phase) enrollment

     1. Untreated AML who cannot tolerate standard induction chemotherapy;
     2. Untreated higher-risk MDS;
* The main organs function well.
* Subjects must be willing to provide available diagnostic evidence or perform bone marrow aspiration and biopsy before the study treatment and must be willing to perform bone marrow aspiration and biopsy after receiving the study treatment.
* Female subjects of childbearing age should agree to use contraceptive measures (such as intrauterine devices, contraceptives or condoms) during the study period and within 6 months after the end of the study; negative serum pregnancy test within 7 days before study enrollment, and must be non-lactating subjects; male subjects should agree to use contraceptive measures during the study period and within 6 months after the end of the study period.

Exclusion Criteria:

* Tumor disease and medical history:

  1. central nervous system leukemia;
  2. Other malignant tumors have occurred or are currently suffering from other malignant tumors within 3 years. The following two conditions can be included: other malignancies treated by a single surgery, achieving 5 years of continuous disease-free survival (DFS);
  3. Clinically significant uncontrolled pleural effusion, ascites, moderate or more remarkable pericardial effusion requiring repeated drainage.
* Previous anti-tumor therapy:

  1. Previous use of other drugs targeting the CD47/signal-regulatory protein α (SIRPα) signaling pathway;
  2. Received any antibody drug treatment under investigation within 4 weeks before the first administration, received Chimeric Antigen Receptor -T (CAR-T) therapy, or other immune cell therapy, or autologous hematopoietic stem cell transplantation 3 months before the first administration;
  3. Previously received allogeneic hematopoietic stem cell transplantation;
  4. Received any major surgery, chemotherapy and/or radiotherapy, immunotherapy or targeted therapy within 4 weeks before the first administration;
  5. The first administration is less than 5 drug half-lives from the previous oral targeted therapy (calculated from the end of the last treatment);
  6. Received Chinese patent medicines with anti-tumor indications within 2 weeks before the first administration, including compound mylabris capsules, Kangai injection, Kanglaite capsule/injection, Aidi injection, javanica oil, Xiao'ai ping tablet/injection, cinobufagin capsule, etc., (using symptomatic treatment such as hydroxyurea, leukocyte apheresis and erythropoietin and other hematopoietic growth factors within 7 days is allowed);
* Combined diseases and medical history:

  1. Liver abnormalities:

     1. Decompensated cirrhosis (Child-Pugh liver function grade B or C);
     2. Hepatitis B virus infection;
     3. Hepatitis C virus infection;
  2. Kidney abnormalities:

     1. Renal failure requires hemodialysis or peritoneal dialysis;
     2. history of nephrotic syndrome.
  3. Gastrointestinal abnormalities:

     1. Persistent chronic diarrhea despite maximal medical treatment;
     2. Active inflammatory bowel disease (such as ulcerative colitis, Crohn's disease) within 4 weeks before the first dose.
  4. Cardiovascular and cerebrovascular abnormalities:

     1. Concomitant or previous history of central nervous system disease, including seizures, hemorrhagic/ischemic stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disease, paralysis, aphasia, mental illness, disturbance of consciousness, unknown Cause coma, neuropathy, organic brain syndrome, etc.;
     2. Brain Magnetic Resonance Imaging (MRI) evidence of inflammatory lesions and/or vasculitis;
     3. Cerebrovascular accident, cerebral infarction, etc., occurred within 6 months before the first administration;
     4. Arterial/venous thrombosis events such as deep vein thrombosis and pulmonary embolism occurred within 6 months before the first administration;
     5. Accompanying or previous history of cardiovascular disease, including grade III or IV heart failure defined by the New York Heart Association classification, atrioventricular block of grade II and above, myocardial infarction within 6 months before the first dose, severe History of arrhythmia, unstable angina, etc.;
     6. Hypertension that cannot be controlled by the combination of two drugs (at least 2 measurements are systolic blood pressure ≥ 160 mmHg, diastolic blood pressure ≥ 100 mmHg);
     7. Previously or currently suffering from heart valvulitis and endarteritis.
  5. History of immunodeficiency:

     1. Known human immunodeficiency virus (HIV) infection or other acquired or congenital immunodeficiency diseases;
     2. Prepare to undergo or have previously received organ transplantation or have noticeable host transplantation reactions;
     3. Need to receive systemic immunosuppressant therapy, including but not limited to the use of cyclosporine, tacrolimus, etc., within 4 weeks before the first administration, and receive high-dose glucocorticoid therapy (prednisone >30 mg /day or other glucocorticoids at equivalent doses), or those with autoimmune diseases, allergic diseases or immune rejection receiving any other immunosuppressive therapy. Patients receiving inhaled or topical corticosteroids or prednisone < 10 mg/day or equivalent doses of other systemic corticosteroids at a stable dose for at least 4 weeks before the first dose or receiving Prophylactic medication to prevent infusion reactions can be selected.
  6. Uncontrolled active systemic bacterial, fungal, or viral infection.
  7. Unexplained fever > 38.5 ℃ occurred during screening or before the first medication (except for fever caused by tumors judged by the investigator).
  8. Subjects with any history of hemolytic anemia (including Evans syndrome) or positive Coombs test within 3 months before the first administration.
  9. Lung disease:

     1. Blood oxygen saturation ≤ 95% at rest;
     2. Previous or current noninfectious pneumonia requiring corticosteroid therapy (including but not limited to acute respiratory distress syndrome, acute hypersensitivity pneumonia, drug-associated pneumonia, bronchospasm, acute interstitial pneumonia, idiopathic pulmonary interstitial fibrosis, etc.);
     3. Evidence of active pneumonia found on chest Computed Tomography (CT) scan during the screening period;
     4. Active tuberculosis.
  10. A history of severe allergies of unknown causes; known allergies to monoclonal antibody drugs or exogenous human immunoglobulins; known allergies to study drug excipients.
  11. Combined with serious or not well-controlled concomitant diseases that, according to the investigator's judgment, seriously endanger the subject's safety or affect the study's completion.
  12. With or previous history of pituitary or adrenal dysfunction (as assessed by the investigator).
  13. History of drug abuse or drug abuse.
  14. myelodysplastic syndromes (MDS) subjects combined with the following two conditions: uncorrected folic acid and vitamin B12 deficiency MDS transformed from pre-existing myeloproliferative neoplasms (MPN) or MDS/MPN types that meet the World Health Organization (WHO) 2016 classification criteria, including chronic Myeloid leukemia (CMML), atypical chronic myeloid leukemia (CML), juvenile myeloid leukemia (JMML).
  15. M3 type acute myeloid leukemia (AML) and AML with positive BCR-ABL mutation gene.
* Inoculation within 4 weeks before the first administration or vaccination with live attenuated vaccine during the planned study period.
* Participated in other drug clinical trials within the past 30 days.
* It is estimated that the compliance of patients participating in this clinical research needs to be improved.
* Hypersensitivity to azacitidine or mannitol;

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | Up to 2 years.
  Adverse events refer to all adverse medical events that occur after patients receive the experimental drug, which can be manifested as symptoms, signs, diseases or abnormal laboratory tests, but do not necessarily have a causal relationship with the experimental drug. Evaluated by Common Terminology Criteria for Adverse Events 5.0 (CTCAE 5.0).
Incidence of serious adverse events (SAEs) | Up to 2 years.
  Incidence of serious adverse events (SAEs) evaluated by CTCAE 5.0.
Severity of serious adverse events (SAEs) | Up to 2 years.
  Severity of serious adverse events (SAEs) evaluated by CTCAE 5.0.

SECONDARY OUTCOMES:
The area under the curve (AUC) | Day1 and Day 22 of Cycle 1: pre-dose, 5 min, 2 h, 6 h, 24 h, 72 h, 120 hours after dose; Cycle 1 Day 8, Cycle 1 Day 15, Cycle 2 Day 1, Cycle 2 Day 15: pre-dose, 5 min after dose; 90 days after last dose; Each cycle is 28 days.
  The area under the curve (AUC) of serum or plasma concentration of TQB2928
Peak concentration (Cmax) | Day1 and Day 22 of Cycle 1: pre-dose, 5 min, 2 h, 6 h, 24 h, 72 h, 120 hours after dose; Cycle 1 Day 8, Cycle 1 Day 15, Cycle 2 Day 1, Cycle 2 Day 15: pre-dose, 5 min after dose; 90 days after last dose; Each cycle is 28 days.
  Maximum observed concentration of TQB2928
Peak Time (Tmax) | Day1 and Day 22 of Cycle 1: pre-dose, 5 min, 2 h, 6 h, 24 h, 72 h, 120 hours after dose; Cycle 1 Day 8, Cycle 1 Day 15, Cycle 2 Day 1, Cycle 2 Day 15: pre-dose, 5 min after dose; 90 days after last dose; Each cycle is 28 days.
  Time to reach maximum concentration of TQB2928
Incidence of anti-drug antibody (ADA) | Cycle1 Day1 and Cycle 5 Day 1: pre-dose, 5 min, 2 h, 6 h, 24 h, 72 h, 120 hours after dose; 90 days after last dose; Each cycle is 28 days.
  Incidence of anti-drug antibody (ADA)
AML: Objective Response Rate (ORR) | Up to 2 years.
  Defined as the percentage of Complete Response (CR) plus partial response (PR) plus Complete Response with incomplete hematological recovery (CRi) plus Morphological absence of leukemia status (MLFS) plus Complete Response with incomplete hematological recovery (CRh)
AML: Duration of Response (DOR) | Up to 2 years.
  For all patients with a best response of CR, CRh, CRi, MLFS, or PR, the time from the date of first achieved remission to the date of first documented disease progression/relapse/treatment failure or death, whichever occurs first.
AML: Time to CR+CRh+CRi | Up to 2 years.
  The time from the date of first TQB2928 injection treatment to the date of first CR, CRh or CRi among all patients whose best response was CR, CRh or CRi.
AML: Event-free survival (EFS) | Up to 2 years.
  Refers to the time from the date of receiving the first TQB2928 injection treatment to the first clearly recorded date of recurrence after remission, disease progression/treatment failure or death, whichever occurs first.
AML: Relapse-Free Survival (RFS) | Up to 2 years.
  Refers to the time from the date of remission to the first clearly recorded hematological relapse or death from any cause for patients who have achieved CR, CRh, or CRi, whichever occurs first.
AML: Overall survival (OS) | Up to 2 years.
  The time from the date of receiving the first TQB2928 injection treatment to the date of death from any cause.
MDS: Complete Response (CR) Rate | Up to 2 years.
  Proportion of patients whose best response is Complete Response
MDS: Objective Response Rate (ORR) | Up to 2 years.
  Proportion of patients with best response in CR, Complete molecular remission (mCR), PR or hematological remission
MDS: Improvement in Transfusion Independence | Up to 2 years.
  Proportion of patients who were transfusion dependent at baseline who were free of red-blood-cell (RBC)/platelet transfusion after first dose.
MDS: Progression Free Survival (PFS) | Up to 2 years.
  From the date of receiving the first TQB2928 injection treatment to the first documented time to investigator-assessed disease progression/relapse after CR or death from any cause.
MDS: Leukemia-free survival | Up to 2 years.
  From the date of receiving the first TQB2928 injection treatment to the blast cells in bone marrow/peripheral blood exceeding 20%, or the time of diagnosis of extramedullary acute leukemia, or death due to any cause.
MDS: Change from Baseline in Quality of Life (QoL) Score | Up to 2 years.
  Proportion of patients with a confirmed improvement of at least 10 points from baseline in overall health status/ QoL score assessed using the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-C30 (QLQ-C30)
MDS: Change from Baseline in the Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue | Up to 2 years.
  Proportion of patients with confirmed improvement of at least 3 points from baseline in FACIT-Fatigue score

CONTACTS AND LOCATIONS:
Locations (9):
- China (9):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Chongqing Hospital of Traditional Chinese Medicine, Chongqing, Chongqing Municipality
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Shanghai Jiaotong University, School of Medicine, Ruijin Hospital, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang